CLINICAL TRIAL: NCT04026412
Title: A Phase 3, Randomized, Open Label Study to Compare Nivolumab Plus Concurrent Chemoradiotherapy (CCRT) Followed by Nivolumab Plus Ipilimumab or Nivolumab Plus CCRT Followed by Nivolumab vs CCRT Followed by Durvalumab in Previously Untreated, Locally Advanced Non-small Cell Lung Cancer (LA NSCLC)
Brief Title: A Study of Nivolumab and Ipilimumab in Untreated Participants With Stage 3 Non-small Cell Lung Cancer (NSCLC) That is Unable or Not Planned to be Removed by Surgery
Acronym: CheckMate73L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-73L; 2019-001222-98 (EudraCT Number)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: nivolumab + CCRT + ipilimumab (Experimental): Concurrent chemoradiotherapy (CCRT)
  Interventions: Biological: nivolumab; Biological: ipilimumab
- Arm B: nivolumab + CCRT (Experimental): Concurrent chemoradiotherapy (CCRT)
  Interventions: Biological: nivolumab
- Arm C: CCRT + durvalumab (Experimental): Concurrent chemoradiotherapy (CCRT)
  Interventions: Biological: durvalumab

INTERVENTIONS:
Biological: nivolumab — Specified dose on specified days
  Arms: Arm A: nivolumab + CCRT + ipilimumab; Arm B: nivolumab + CCRT
Biological: ipilimumab — Specified dose on specified days
  Arms: Arm A: nivolumab + CCRT + ipilimumab
Biological: durvalumab — Specified dose on specified days
  Arms: Arm C: CCRT + durvalumab

SUMMARY:
The primary purpose of the study is to compare the effectiveness of nivolumab plus concurrent chemoradiotherapy (CCRT) followed by nivolumab plus ipilimumab vs CCRT followed by durvalumab in participants with untreated Locally Advanced Non-small Cell Lung Cancer (LA NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Locally advanced stage IIIA, IIIB, or IIIC (T1-2 N2-3 M0, T3 N1-3 M0, or T4 N0-3 M0) pathologically-confirmed NSCLC, according to 8th TNM classification. Participants who are not planned for potential curative surgical resection are eligible.
* Newly diagnosed and treatment-naïve, with no prior local or systemic anticancer therapy given as primary therapy for locally advanced disease

Exclusion Criteria:

* Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator would preclude the participant from adhering to the protocol or would increase the risk associated with study participation
* Active infection requiring systemic therapy within 14 days prior to randomization
* History of organ or tissue transplant that requires systemic use of immune suppressive agents
* Prior thoracic radiotherapy

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (181):
- United States (24):
  - Local Institution - 0119, La Jolla, California
  - Local Institution - 0207, San Francisco, California
  - Local Institution - 0166, San Francisco, California
  - Local Institution - 0129, Lone Tree, Colorado
  - Local Institution - 0233, Jacksonville, Florida
  - Local Institution - 0219, Orlando, Florida
  - Local Institution - 0039, Pensacola, Florida
  - Local Institution - 0125, Atlanta, Georgia
  - Local Institution - 0165, Augusta, Georgia
  - Local Institution - 0218, Edgewood, Kentucky
  - Local Institution - 0108, Bethesda, Maryland
  - Local Institution - 0116, Traverse City, Michigan
  - Local Institution - 0053, Cincinnati, Ohio
  - Local Institution - 0131, Cincinnati, Ohio
  - Local Institution - 0188, Cincinnati, Ohio
  - Local Institution - 0112, Cleveland, Ohio
  - Local Institution - 0124, Cleveland, Ohio
  - Local Institution - 0047, Cleveland, Ohio
  - Local Institution - 0123, Youngstown, Ohio
  - Local Institution - 0077, Charleston, South Carolina
  - Local Institution - 0191, Austin, Texas
  - Local Institution - 0079, Bryan, Texas
  - Local Institution - 0130, Dallas, Texas
  - Local Institution - 0071, Burlington, Vermont
- Argentina (4):
  - Local Institution - 0044, CABA, Buenos Aires
  - Local Institution - 0045, Río Cuarto, Córdoba Province
  - Local Institution - 0043, Buenos Aires, Distrito Federal
  - Local Institution - 0042, Caba, Distrito Federal
- Australia (9):
  - Local Institution - 0031, Darlinghurst, New South Wales
  - Local Institution - 0134, Gosford, New South Wales
  - Local Institution - 0033, Kingswood, New South Wales
  - Local Institution - 0029, Greenslopes, Queensland
  - Local Institution - 0028, Adelaide, South Australia
  - Local Institution - 0224, Ballarat Central, Victoria
  - Local Institution - 0052, Melbourne, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution - 0030, Murdoch, Western Australia
- Belgium (4):
  - Local Institution - 0003, Brussels
  - Local Institution - 0001, Ghent
  - Local Institution - 0004, Liège
  - Local Institution - 0002, Yvoir
- Brazil (6):
  - Local Institution - 0038, Ipatinga, Minas Gerais
  - Local Institution - 0234, Ijuí, Rio Grande do Sul
  - Local Institution - 0034, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0037, Blumenau, Santa Catarina
  - Local Institution - 0036, Barretos, São Paulo
  - Local Institution - 0035, Rio de Janeiro
- Canada (6):
  - Local Institution - 0127, Kingston, Ontario
  - Local Institution - 0078, Oshawa, Ontario
  - Local Institution - 0237, Chicoutimi, Quebec
  - Local Institution - 0126, Québec, Quebec
  - Local Institution - 0070, Rimouski, Quebec
  - Local Institution - 0092, Trois-Rivières, Quebec
- Chile (2):
  - Local Institution - 0040, Viña del Mar, Región de Valparaíso
  - Local Institution - 0041, Santiago, Santiago Metropolitan
- China (20):
  - Local Institution - 0146, Beijing, BEI
  - Local Institution - 0149, Chongqing, Chongqing Municipality
  - Local Institution - 0179, Fuzhou, Fujian
  - Local Institution - 0164, Xiamen, Fujian
  - Local Institution - 0192, Guiyang, Guizhou
  - Local Institution - 0147, Hankou, Hubei
  - Local Institution - 0148, Wuhan, Hubei
  - Local Institution - 0150, Wuhan, Hubei
  - Local Institution - 0154, Changsha, Hunan
  - Local Institution - 0139, Nanjing, Jiangsu
  - Local Institution - 0178, Nanchang, Jiangxi
  - Local Institution - 0170, Changchun, Jilin
  - Local Institution - 0183, Changchun, Jilin
  - Local Institution - 0180, Gongzhuling, Jilin
  - Local Institution - 0138, Jinan, Shandong
  - Local Institution - 0145, Shanghai, Shanghai Municipality
  - Local Institution - 0186, Chengdu, Sichuan
  - Local Institution - 0189, Chengdu, Sichuan
  - Local Institution - 0140, Hangzhou, Zhejiang
  - Local Institution - 0184, Linhai, Zhejiang
- France (10):
  - Local Institution - 0086, Bordeaux
  - Local Institution - 0087, Dijon
  - Local Institution - 0081, Lyon
  - Local Institution - 0082, Montpellier
  - Local Institution - 0084, Nantes
  - Local Institution - 0227, Paris
  - Local Institution - 0091, Paris
  - Local Institution - 0083, Paris
  - Local Institution - 0090, Paris
  - Local Institution - 0089, Tours
- Germany (10):
  - Local Institution - 0060, Berlin
  - Local Institution - 0063, Essen
  - Local Institution - 0076, Großhansdorf
  - Local Institution - 0101, Hamm
  - Local Institution - 0073, Heidelberg
  - Local Institution - 0061, Immenhausen
  - Local Institution - 0062, Kempten
  - Local Institution - 0075, Löwenstein
  - Local Institution - 0109, Mainz
  - Local Institution - 0072, Stuttgart
- Greece (4):
  - Local Institution - 0161, Athens
  - Local Institution - 0135, Athens
  - Local Institution - 0136, Larissa
  - Local Institution - 0162, N.Kifissia
- Ireland (2):
  - Local Institution - 0024, Dublin, Dublin
  - Local Institution - 0023, Dublin
- Italy (7):
  - Local Institution - 0114, Monza (MB), Monza (MB)
  - Local Institution - 0068, Brescia
  - Aou Policlinico V. Emanuele Di Catania, Catania
  - Azienda Ospedaliero-Universitaria Mater Domini, Catanzaro
  - Local Institution - 0050, Lucca
  - Local Institution - 0115, Milan
  - Local Institution - 0048, Perugia
- Japan (20):
  - Local Institution - 0204, Nagoya, Aichi-ken
  - Local Institution - 0212, Fukuoka, Fukuoka
  - Local Institution - 0211, Kurume-shi, Fukuoka
  - Local Institution - 0197, Ōta, Gunma
  - Local Institution - 0195, Sapporo, Hokkaido
  - Local Institution - 0206, Kobe, Hyōgo
  - Local Institution - 0203, Kanazawa, Ishikawa-ken
  - Local Institution - 0216, Yokohama, Kanagawa
  - Local Institution - 0201, Yokohama, Kanagawa
  - Local Institution - 0217, Yokohama, Kanagawa
  - Local Institution - 0196, Sendai, Miyagi
  - Local Institution - 0202, Niigata, Niigata
  - Local Institution - 0205, Osaka, Osaka
  - Local Institution - 0210, Sayama, Osaka
  - Local Institution - 0198, Hidaka-shi, Saitama
  - Local Institution - 0174, Kitaadachi-gun, Saitama
  - Local Institution - 0199, Bunkyo-ku, Tokyo
  - Local Institution - 0200, Chuo-ku, Tokyo
  - Local Institution - 0232, Ube, Yamaguchi
  - Local Institution - 0175, Wakayama
- Mexico (5):
  - Local Institution - 0027, La Paz, BAJA Californa SUR
  - Local Institution - 0080, Guadalajara, Jalisco
  - Local Institution - 0067, Df, Mexico City
  - Local Institution - 0014, Monterrey, Nuevo León
  - Local Institution - 0015, Culiacán, Sinaloa
- Netherlands (5):
  - Local Institution - 0006, Amsterdam
  - Local Institution - 0025, Arnhem
  - Local Institution - 0240, Leiden
  - Local Institution - 0005, Maastrict
  - Local Institution - 0026, Veldhoven
- Poland (4):
  - Local Institution - 0107, Bydgoszcz
  - Local Institution - 0102, Gdansk
  - Local Institution - 0104, Krakow
  - Local Institution - 0235, Tomaszów Mazowiecki
- Puerto Rico (2):
  - Local Institution - 0120, Hato Rey
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- Romania (6):
  - Local Institution - 0018, Bucharest
  - Local Institution - 0222, Bucharest
  - Local Institution - 0019, Cluj-Napoca
  - Local Institution - 0020, Constanța
  - Local Institution - 0017, Craiova
  - Local Institution - 0021, Floresti/ Cluj
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution - 0171, Singapore, Singapore
- South Korea (3):
  - Local Institution - 0167, Cheongju-si, Chungcheonbuk-do,
  - Local Institution - 0152, Seoul
  - Local Institution - 0168, Seoul
- Spain (8):
  - Local Institution - 0106, Barcelona
  - Local Institution - 0099, L'Hospitalet de Llobregat
  - Local Institution - 0096, Madrid
  - Local Institution - 0095, Madrid
  - Local Institution - 0098, Pamplona
  - Local Institution - 0105, Santiago de Compostela
  - Local Institution - 0097, Seville
  - Local Institution - 0100, Zaragoza
- Sweden (2):
  - Local Institution - 0065, Gothenburg, Västra Götaland County
  - Local Institution - 0064, Stockholm
- Switzerland (4):
  - Local Institution - 0057, Basel
  - Local Institution - 0058, Lausanne
  - Local Institution - 0059, Sankt Gallen
  - Local Institution - 0056, Zurich
- Taiwan (6):
  - Local Institution - 0208, KaohsiungCity
  - Local Institution - 0214, New Taipei City
  - Local Institution - 0209, Tainan
  - Local Institution - 0213, Taipei
  - Local Institution - 0133, Taipei
  - Local Institution - 0143, Taipei
- United Kingdom (5):
  - Local Institution - 0010, Poole, Dorset
  - Local Institution - 0012, Swansea, Glamorgan
  - Local Institution - 0054, Aberdeen
  - Local Institution - 0007, Bebington
  - Local Institution - 0009, Hull

REFERENCES:
- [Derived] De Ruysscher D, Ramalingam S, Urbanic J, Gerber DE, Tan DSW, Cai J, Li A, Peters S. CheckMate 73L: A Phase 3 Study Comparing Nivolumab Plus Concurrent Chemoradiotherapy Followed by Nivolumab With or Without Ipilimumab Versus Concurrent Chemoradiotherapy Followed by Durvalumab for Previously Untreated, Locally Advanced Stage III Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2022 May;23(3):e264-e268. doi: 10.1016/j.cllc.2021.07.005. Epub 2021 Jul 19. PMID 34489161
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A:Nivo + CCRT/Nivo + Ipi: Participants with Previously Untreated, Locally Advanced Non-small Cell Lung Cancer (LA NSCLC) received intravenous infusion of 360 mg Nivolumab once in 3 weeks (Q3W) Plus concurrent chemoradiotherapy (CCRT) Q3W up to 3 cycles (each cycle of 21 days) followed by recovery of 42 days followed by maintenance treatment of intravenous infusion Nivolumab 360 mg Q3W plus Ipilimumab 1 mg/kg Q6W for up to 1 year.
- Arm B: Nivo + CCRT/Nivo: Participants with Previously Untreated, Locally Advanced Non-small Cell Lung Cancer (LA NSCLC) received intravenous infusion of 360 mg Nivolumab once in 3 weeks (Q3W) Plus concurrent chemoradiotherapy (CCRT) Q3W up to 3 cycles (each cycle of 21 days) followed by recovery of 42 days followed by maintenance treatment of intravenous infusion Nivolumab 480 mg once in 4 weeks Q4W for up to 1 year.
- Arm C: CCRT/Durva: Participants with Previously Untreated, Locally Advanced Non-small Cell Lung Cancer (LA NSCLC) received CCRT Q3W for up to 3 cycles (each cycle is of 21 days) followed by recovery of 42 days followed by intravenous infusion of Durvalumab 10 mg/kg Q2W for up to 1 year.
Period: Overall Study
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Started | 287 | 320 | 318
Completed | 103 | 138 | 144
Not Completed | 184 | 182 | 174

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva | Total
Number analyzed (Participants) | 287 | 320 | 318 | 925
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.99) | 63.7 (8.50) | 63.9 (9.18) | 63.8 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 76 | 79 | 222
  Male | 220 | 244 | 239 | 703
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 32 | 32 | 92
  Not Hispanic or Latino | 155 | 167 | 157 | 479
  Unknown or Not Reported | 104 | 121 | 129 | 354
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 93 | 119 | 105 | 317
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 2 | 11
  White | 182 | 192 | 204 | 578
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Arm A Vs Arm C - Progression-Free Survival (PFS) by RECIST 1.1 Per Blinded Independent Central Review (BICR)
Description: Progression-Free Survival then (PFS) is defined as the time between the date of randomization and the date of first documented disease progression, based on BICR assessments (per RECIST v1.1), or death due to any cause, whichever occurs first based on Kaplan-Meier estimates. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 53 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study. Participant in Arm A and C were only considered in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 318
months | 16.69 [12.58 to 21.98] | 15.64 [13.67 to 19.75]
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; p = 0.6460, Cox proportional hazards model; Hazard Ratio (HR) = 0.95, 96% CI 2-sided [0.77 to 1.19]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) for all randomized participants is the time between randomization and the date of death from any cause based on Kaplan-Meier estimates. For participants who are alive, their survival time was censored at the last date that they were known to be alive. OS was censored for participants at the date of randomization if they had no follow-up.
Time Frame: From randomization untill death (up to approximately 61 months)
Population: All enrolled participants who are randomized to any treatment arm in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
months | 34.60 [26.81 to NA] — UL for 95% CI Not estimable due to insufficient number of events. | 39.49 [33.48 to NA] — UL for 95% CI Not estimable due to insufficient number of events. | 39.79 [30.92 to NA] — UL for 95% CI Not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.87 to 1.41]
Statistical Analysis 2: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.75 to 1.22]
Statistical Analysis 3: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Hazard Ratio, log = 1.16, 95% CI 2-sided [0.91 to 1.48]

3. Secondary Outcome: Arm B Vs Arm C and Arm A Vs Arm B- Progression-Free Survival (Irrespective of Subsequent Therapy) by RECIST 1.1 Per Blinded Independent Central Review (BICR)
Description: Progression-Free Survival (PFS) is defined as the time between the date of randomization and the date of first documented disease progression, based on BICR assessments (per RECIST v1.1), or death due to any cause, whichever occurs first based on Kaplan-Meier estimates. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
months | 16.82 [12.58 to 22.05] | 17.38 [14.09 to 22.14] | 15.67 [13.77 to 20.83]
Statistical Analysis 1: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.05]
Statistical Analysis 2: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.93 to 1.42]

4. Secondary Outcome: Objective Response Rate (ORR) by BICR
Description: Objective Response Rate (ORR) is defined as the percentage of participants whose best overall response (BOR) is either CR or PR by blinded independent central review (BICR) per response evaluation criteria in solid tumors (RECIST) v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
percentage of participants | 67.6 [61.8 to 73.0] | 72.2 [66.9 to 77.0] | 64.5 [58.9 to 69.7]
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; Difference in ORR = 3.2, 95% CI 2-sided [-4.1 to 10.6]
Statistical Analysis 2: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Difference in ORR = 7.8, 95% CI 2-sided [0.7 to 14.8]
Statistical Analysis 3: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Difference in ORR = -4.7, 95% CI 2-sided [-11.8 to 2.5]

5. Secondary Outcome: Duration of Response (DoR) by RECIST 1.1 Per BICR
Description: Duration of objective response (DoR) is defined as the time between the date of first confirmed response (CR or PR) to the date of the first documented tumor progression (per RECIST 1.1) per BICR assessment, or death due to any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study. Participants with CR or PR were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 194 | 231 | 205
months | 25.76 [2.1 to 47.9] | 31.84 [1.6 to 44.3] | 25.17 [1.0 to 44.3]

6. Secondary Outcome: Time to Response (TTR) by RECIST 1.1 Per BICR
Description: Time to response (TTR) is defined as the time, in months, from randomization to the first objective documentation of PR or better assessed per BICR.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 194 | 231 | 205
months | 2.92 [0.9 to 22.2] | 2.96 [1.3 to 41.9] | 2.92 [1.2 to 24.9]

7. Secondary Outcome: Progression Free Survival (PFS) by RECIST 1.1 Per Investigator Assessment
Description: Progression-Free Survival then (PFS) is defined as the time between the date of randomization and the date of first documented disease progression, based on Investigator assessments (per RECIST v1.1), or death due to any cause, whichever occurs first Calculated using Kaplan-Meier estimates. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
months | 16.82 [13.83 to 20.40] | 17.71 [13.83 to 24.71] | 16.53 [13.77 to 19.38]
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.82 to 1.23]
Statistical Analysis 2: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.05]
Statistical Analysis 3: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.95 to 1.44]

8. Secondary Outcome: Objective Response Rate (ORR) by RECIST 1.1 Per Investigator Assessment
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR by investigator assessment per response evaluation criteria in solid tumors (RECIST) v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
percentage of participants | 61.3 [55.4 to 67.0] | 63.1 [57.6 to 68.4] | 57.9 [52.2 to 63.4]
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; Difference in ORR = 3.5, 95% CI 2-sided [-4.1 to 11.1]
Statistical Analysis 2: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Difference in ORR = 5.4, 95% CI 2-sided [-2.0 to 12.9]
Statistical Analysis 3: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Difference in ORR = -1.9, 95% CI 2-sided [-9.5 to 5.6]

9. Secondary Outcome: Duration of Response (DOR) by RECIST 1.1 Per Investigator Assessment
Description: Duration of objective response (DoR) is defined as the time between the date of first confirmed response (CR or PR) to the date of the first documented tumor progression (per RECIST 1.1) per investigator assessment, or death due to any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 176 | 202 | 184
months | 22.83 [0.0 to 47.4] | 33.18 [0.0 to 47.6] | 27.93 [0.0 to 46.5]

10. Secondary Outcome: Time to Response (TTR) by RECIST 1.1 Per Investigator Assessment
Description: Time to response (TTR) is defined as the time, in months, from randomization to the first objective documentation of PR or better assessed per investigator assessment.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 61 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 176 | 202 | 184
months | 2.96 [1.9 to 25.2] | 2.92 [1.9 to 16.5] | 2.89 [1.4 to 22.1]

11. Secondary Outcome: Time to Death or Distant Metastases (TDDM)
Description: Time to Death or Distant Metastases (TDDM) is defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis based on Kaplan-Meier estimates. Distant metastasis is defined as any new lesion that is outside of the thorax (except for heart) according to RECIST 1.1, as assessed by the Investigator.
Time Frame: From randomization until metastases or death, whichever occurs first (up to approximately 61 months)
Population: Intent-to-Treat population includes all enrolled participants who are randomized to any treatment arm in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 287 | 320 | 318
months | 30.65 [22.57 to NA] — UL of 95% CI not estimable due to insufficient number of events | 36.14 [25.86 to NA] — UL of 95% CI not estimable due to insufficient number of events | 30.36 [21.62 to 40.15]
Statistical Analysis 1: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.23]
Statistical Analysis 2: Comparison: Arm B: Nivo + CCRT/Nivo vs Arm C: CCRT/Durva; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.65 to 1.06]
Statistical Analysis 3: Comparison: Arm A:Nivo + CCRT/Nivo + Ipi vs Arm B: Nivo + CCRT/Nivo; Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.91 to 1.49]

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs and Select AEs
Description: An Adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporarily associated with the use of medicinal product, whether or not considered related to the investigational medicinal product. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose (Day 1) till 30 days after the last dose (up to approximately 19 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 282 | 318 | 317
Participants
  ADVERSE EVENTS | 279 | 315 | 312
  SERIOUS ADVERSE EVENTS | 155 | 156 | 136
  GASTROINTESTINAL ADVERSE EVENT | 67 | 60 | 54
  HEPATIC ADVERSE EVENT | 55 | 59 | 72
  PULMONARY ADVERSE EVENT | 87 | 92 | 55
  RENAL ADVERSE EVENT | 25 | 16 | 32
  SKIN ADVERSE EVENT | 111 | 115 | 115
  HYPERSENSITIVITY/INFUSION REACTION | 18 | 17 | 9

13. Secondary Outcome: Change From Baseline in Non-small Cell Lung Cancer (NSCLC)-Symptom Assessment Questionnaire (SAQ) Total Score at Week 48
Description: The NSCLC-SAQ is a questionnaire used in clinical trials to understand how non-small cell lung cancer (NSCLC) affects your daily life and well-being. It has 7 questions that ask about your symptoms over the past 7 days, including cough, pain, shortness of breath, fatigue, and appetite loss. The total scores from the questionnaire range from 0 to 20. A higher score means you have more severe symptoms and are feeling worse, which is a bad outcome. A lower score means you have fewer symptoms and are feeling better, which is a good outcome.
Time Frame: Baseline (Day 1) and Week 48
Population: All randomized participants. Only participants with data available at the specified timepoint are included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
Number analyzed (Participants) | 83 | 109 | 120
Score on a Scale | -0.60 (3.260) | -0.91 (3.507) | -0.89 (3.731)

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from randomization until death due to any cause (up to approximately 61 months). Serious and Non-serious AEs were collected from first dose (Day 1) till 30 days after the last dose (up to approximately 19 months).
Description: All-cause mortality was collected for intent-to-treat population. Serious and Non-serious AEs were collected for all the treated participants.
Arm/Group | Arm A:Nivo + CCRT/Nivo + Ipi | Arm B: Nivo + CCRT/Nivo | Arm C: CCRT/Durva
All-Cause Mortality (participants affected / at risk) | 132/287 | 132/320 | 132/318
Serious Adverse Events (participants affected / at risk) | 180/282 | 181/318 | 145/317
Other Adverse Events (participants affected / at risk) | 273/282 | 310/318 | 307/317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A:Nivo + CCRT/Nivo + Ipi (N=282) | Arm B: Nivo + CCRT/Nivo (N=318) | Arm C: CCRT/Durva (N=317)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 9
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 2 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 3
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric artery embolism (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 8 | 4
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 2
Chest pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Death (General disorders) | 2 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 3
General physical health deterioration (General disorders) | 1 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1
Medical device site fistula (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 5
Sudden death (General disorders) | 1 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 9 | 11 | 6
COVID-19 pneumonia (Infections and infestations) | 2 | 4 | 5
Cellulitis (Infections and infestations) | 2 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 0
Cytomegalovirus enterocolitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Empyema (Infections and infestations) | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Haematological infection (Infections and infestations) | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 2 | 1 | 3
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Lung abscess (Infections and infestations) | 1 | 1 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0 | 0
Pneumonia (Infections and infestations) | 33 | 39 | 29
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 3 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 3 | 0
Sepsis (Infections and infestations) | 5 | 4 | 1
Septic shock (Infections and infestations) | 2 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 5 | 4 | 4
Radiation pneumonitis (Injury, poisoning and procedural complications) | 18 | 15 | 13
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 1
Granulocyte count decreased (Investigations) | 0 | 0 | 1
Imaging procedure abnormal (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 3
Platelet count decreased (Investigations) | 2 | 2 | 6
White blood cell count decreased (Investigations) | 2 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 12 | 14
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 0
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 13 | 10 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 32 | 32 | 11
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A:Nivo + CCRT/Nivo + Ipi (N=282) | Arm B: Nivo + CCRT/Nivo (N=318) | Arm C: CCRT/Durva (N=317)
Anaemia (Blood and lymphatic system disorders) | 124 | 132 | 134
Leukopenia (Blood and lymphatic system disorders) | 41 | 39 | 46
Lymphopenia (Blood and lymphatic system disorders) | 22 | 25 | 38
Neutropenia (Blood and lymphatic system disorders) | 57 | 62 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 42 | 27 | 29
Hyperthyroidism (Endocrine disorders) | 22 | 16 | 16
Hypothyroidism (Endocrine disorders) | 44 | 51 | 32
Abdominal pain (Gastrointestinal disorders) | 20 | 10 | 17
Abdominal pain upper (Gastrointestinal disorders) | 8 | 17 | 13
Constipation (Gastrointestinal disorders) | 82 | 78 | 89
Diarrhoea (Gastrointestinal disorders) | 64 | 62 | 52
Dyspepsia (Gastrointestinal disorders) | 24 | 21 | 13
Dysphagia (Gastrointestinal disorders) | 53 | 42 | 34
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 5 | 19
Nausea (Gastrointestinal disorders) | 98 | 104 | 108
Odynophagia (Gastrointestinal disorders) | 15 | 20 | 13
Oesophagitis (Gastrointestinal disorders) | 74 | 81 | 69
Vomiting (Gastrointestinal disorders) | 33 | 38 | 31
Asthenia (General disorders) | 60 | 50 | 54
Chest pain (General disorders) | 12 | 11 | 24
Fatigue (General disorders) | 60 | 61 | 77
Non-cardiac chest pain (General disorders) | 19 | 20 | 19
Oedema peripheral (General disorders) | 20 | 20 | 12
Pain (General disorders) | 11 | 13 | 18
Pyrexia (General disorders) | 59 | 46 | 41
COVID-19 (Infections and infestations) | 29 | 41 | 39
Pneumonia (Infections and infestations) | 41 | 43 | 34
Upper respiratory tract infection (Infections and infestations) | 11 | 9 | 17
Radiation oesophagitis (Injury, poisoning and procedural complications) | 48 | 47 | 56
Radiation pneumonitis (Injury, poisoning and procedural complications) | 41 | 52 | 48
Radiation skin injury (Injury, poisoning and procedural complications) | 35 | 46 | 32
Alanine aminotransferase increased (Investigations) | 36 | 35 | 43
Aspartate aminotransferase increased (Investigations) | 26 | 29 | 37
Blood creatine phosphokinase increased (Investigations) | 14 | 20 | 25
Blood creatinine increased (Investigations) | 23 | 13 | 26
Blood thyroid stimulating hormone increased (Investigations) | 9 | 17 | 14
Lymphocyte count decreased (Investigations) | 26 | 42 | 23
Neutrophil count decreased (Investigations) | 54 | 69 | 57
Platelet count decreased (Investigations) | 47 | 55 | 48
Weight decreased (Investigations) | 25 | 24 | 17
White blood cell count decreased (Investigations) | 65 | 73 | 63
Decreased appetite (Metabolism and nutrition disorders) | 79 | 64 | 77
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 21 | 21
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 | 26 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 21 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 29 | 38 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 38 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 26 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 20 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 14 | 23
Dizziness (Nervous system disorders) | 14 | 18 | 12
Headache (Nervous system disorders) | 32 | 30 | 32
Neuropathy peripheral (Nervous system disorders) | 12 | 13 | 16
Insomnia (Psychiatric disorders) | 35 | 37 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 82 | 83 | 87
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 63 | 54
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 17 | 18
Hiccups (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 62 | 76 | 48
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 54 | 69 | 54
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 13 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 65 | 54 | 51
Rash (Skin and subcutaneous tissue disorders) | 51 | 55 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT04026412/Prot_SAP_000.pdf